CLINICAL TRIAL: NCT06911164
Title: Translation, Cultural Adaptation, Reliability, and Validity of the Turkish Version of the Low Back Pain Knowledge Questionnaire
Brief Title: Measurement Properties of the Turkish Version of the Low Back Pain Knowledge Questionnaire
Acronym: LKQ
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Elif AYGUN POLAT, Principal Investigator, Ordu University
Other Study IDs: ODU-SBFTR-AYGUNPOLAT-005; 2024/163 (Other: Ordu University Ethics Committee)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain; Knowledge, Attitudes, Practice
Keywords: reliability; validity
MeSH Terms: conditions — Low Back Pain; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the validity and reliability of the Turkish version of the Low Back Pain Knowledge Questionnaire (LKQ). This questionnaire is a comprehensive, disease-specific tool that evaluates knowledge about low back pain. Adapting it into Turkish will provide healthcare professionals with a valuable resource for assessing patient awareness, guiding educational programs, and improving clinical practices for low back pain management.

DETAILED DESCRIPTION:
This study aims to evaluate the validity and reliability of the Turkish version of the Low Back Pain Knowledge Questionnaire (LKQ), a comprehensive tool that assesses individuals' knowledge about the characteristics, symptoms, causes, and management of low back pain. The study will follow a systematic process, including translation, cultural adaptation, and psychometric evaluation. After translating the questionnaire using the forward-backward method, a panel of experts will review it for clarity and cultural relevance. The adapted questionnaire will be tested on a diverse sample to assess internal consistency (Cronbach's alpha) and test-retest reliability. The results will provide a validated Turkish version of the LKQ, enabling healthcare professionals to assess patient knowledge, guide educational programs, and improve low back pain management and prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or over
* Turkish as their mother tongue
* Presence of back pain of any duration
* Volunteered to participate in the study

Exclusion Criteria:

* Failure to complete the questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low back pain
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-10-04 (Actual)

PRIMARY OUTCOMES:
Low Back Pain Knowledge Questionnaire (LKQ) | first day
  The original LKQ is composed of 16 questions across three dimensions: general knowledge about low back pain (Questions 1, 6, 7, 8, 15), concepts (Questions 2, 3, 4, 5), and treatment (Questions 9, 10, 11, 12, 13, 14, 16). The total score is 24 points, with 8 single-choice questions and 8 multiple-choice questions. Each question has five options, and one point is awarded for each correct answer. A higher total score indicates a greater level of knowledge about low back pain.
Back Beliefs Questionnaire | first day
  The Back Beliefs Questionnaire consists of 14 items to be completed by patients. Nine of these items (Questions 1, 2, 3, 6, 8, 10, 12, 13, 14) are used to assess feelings of helplessness, while the remaining five items (Questions 4, 5, 7, 9, 11) serve as distractors. All items are rated using a 5-point Likert scale, with responses ranging from "1-Strongly Disagree" to "5-Strongly Agree." Scoring is performed by reversing the numerical values selected by the participants and calculating the score based on the helplessness-related items.
Numerical Rating Scale for Pain | first day
  This scale quantitatively assesses pain intensity and is highly sensitive, allowing for easy comparison with other pain scales. Patients are asked to rate their pain severity by selecting a number between 0 and 10.
Roland-Morris Disability Questionnaire | first day
  The Roland-Morris Disability Questionnaire consists of 24 statements that assess an individual's perception of their low back pain and related disabilities. These statements cover areas such as physical functioning/effectiveness (15 items), sleep/rest (3 items), psychosocial issues (2 items), household management (2 items), eating (1 item), and pain frequency (1 item). Each statement is presented to the participant, who is asked to indicate whether it applies to their condition for that day. Scoring is based on the total number of "Yes" responses in the "Yes/No" boxes. As a result, the score can range from 0 (no disability) to 24 (maximum disability).
Low Back Pain Knowledge Questionnaire (LKQ) | 7 days after
  The original LKQ is composed of 16 questions across three dimensions: general knowledge about low back pain (Questions 1, 6, 7, 8, 15), concepts (Questions 2, 3, 4, 5), and treatment (Questions 9, 10, 11, 12, 13, 14, 16). The total score is 24 points, with 8 single-choice questions and 8 multiple-choice questions. Each question has five options, and one point is awarded for each correct answer. A higher total score indicates a greater level of knowledge about low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Elif AYGUN POLAT, PhD, Principal Investigator — Ordu University
Locations (1):
- Ordu university, Altinordu, Ordu, Turkey (Türkiye)